CLINICAL TRIAL: NCT02617186
Title: Robotic Lobectomy vs. Thoracoscopic Lobectomy for Early Stage Lung Cancer: A Randomized Controlled Trial
Brief Title: Robotic Lobectomy vs. Thoracoscopic Lobectomy for Early Stage Lung Cancer: RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: University of Toronto / Toronto General Hospital (Unknown); University of Florida (Other); University Hospital, Rouen (Other); St Vincent's Hospital Melbourne (Other); University of Melbourne / St. Vincent's Private Hospital (Fitzroy, Australia) (Unknown); University of Melbourne / Barwon Health (Geelong, Australia) (Unknown)
Responsible Party: Principal Investigator, Wael Hanna, Associate Professor, Departments of Surgery and HEI, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BFCRS-RP-003-1508-31
Record Dates: First submitted 2015-09-22; First posted 2015-11-30 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer; Thoracic Surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracoscopic Lobectomy (Active Comparator)
  Interventions: Procedure: Video-assisted thoracoscopic surgery
- Robotic Lobectomy (Active Comparator)
  Interventions: Procedure: Robotic thoracic surgery

INTERVENTIONS:
Procedure: Video-assisted thoracoscopic surgery — patients randomized to this arm will receive video-assisted thoracic surgery (VATS)
  Arms: Thoracoscopic Lobectomy
Procedure: Robotic thoracic surgery — patients randomized to this arm will receive robotic thoracic surgery (RTS) with the da Vinci Robot
  Arms: Robotic Lobectomy

SUMMARY:
During video-assisted thoracoscopic lobectomy (VATS), the surgeon inserts a small camera attached to a thoracoscope that puts the image onto a video screen. Instruments are inserted via small incisions, and the lung resection is completed. Robotic thoracic surgery (RTS) uses a similar minimally invasive approach, but the very precise instruments involved with RTS allow the surgeon to view the lung using 3-dimensional imaging. The instruments give the surgeons increased range of motion during the surgery, and research demonstrates that RTS has a less steep learning curve as compared to VATS. Both VATS and RTS demonstrated better results as compared to traditional thoracotomy (open surgery). However, Robotic lobectomy has not yet been compared directly to video-assisted thoracoscopic lobectomy (VATS) in a prospective manner.

There are two major barriers against the widespread adoption of robotic thoracic surgery. The first barrier is the lack of high-quality prospective data. To our knowledge, there are no prospective trials comparing VATS to RTS for early stage lung cancer. The second major barrier to the widespread adoption of robotic technology in thoracic surgery is the perceived higher cost of Robotic lobectomy. To address these barriers, the investigators will undertake the first randomized controlled trial comparing Thoracoscopic Lobectomy to Robotic Lobectomy for early stage lung cancer.

Prospective randomization will eliminate the biases of retrospective data and will serve to determine whether there exist any advantages to Health Related Quality of life (HRQOL) or patient outcomes in favour of Robotic Lobectomy over VATS Lobectomy. Furthermore, through a prospective cost-utility analysis, this trial will provide the highest quality data to evaluate the true economic impact of robotic technology in thoracic surgery in a Canadian health system.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years
2. Clinical stage I, II or IIIa non-small cell lung cancer (NSCLC)
3. Candidates for minimally invasive pulmonary lobectomy, as determined by the operating surgeon.

Exclusion Criteria:

1. Clinical stage IIIb or IV NSCLC
2. Not a candidate for minimally invasive surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2016-01; Primary Completion 2021-09 (Actual); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Difference in HRQOL scores at week 12 between the treatment groups | 12 weeks post-surgery
  Difference in HRQOL scores between the treatment groups, as measured by the EQ-5D-5L questionnaire at week 12.

SECONDARY OUTCOMES:
Short-term clinical outcome differences | 3 weeks post-surgery
  Clinical staging will be determined from diagnostic imaging reports
Short-term clinical outcome differences | 3 weeks post-surgery
  Pathological staging will be determined from pathology report
Short-term clinical outcome differences | 3 weeks post-surgery
  Number of lymph nodes sampled
Short-term clinical outcome differences | 3 weeks post-surgery
  Admission date
Short-term clinical outcome differences | 3 weeks post-surgery
  Date of surgery
Short-term clinical outcome differences | 3 weeks post-surgery
  Discharge date
Short-term clinical outcome differences | 3 weeks post-surgery
  Chest tube removal date
Short-term clinical outcome differences | 3 weeks post-surgery
  Intraoperative blood loss
Short-term clinical outcome differences | 3 weeks post-surgery
  Post-operative analgesia will be determined from list of prescribed pain medications
Short-term clinical outcome differences | 3 weeks post-surgery
  Post-surgical pain will be determined from the Numeric Pain Rating Scale
Resource utilization | 1 year post-surgery
  Operating room time
Resource utilization | 1 year post-surgery
  Operating room staff
Resource utilization | 1 year post-surgery
  Surgical instruments and consumables
Resource utilization | 1 year post-surgery
  Admission to critical care beds
Resource utilization | 1 year post-surgery
  Hospital length of stay
Resource utilization | 1 year post-surgery
  Duration of intravenous analgesia
Resource utilization | 1 year post-surgery
  Postoperative complications
Resource utilization | 1 year post-surgery
  Costs associated with chronic post-surgical pain up to one year after surgery.
Cost Effectiveness | 5 years post-surgery
  The incremental cost per quality-adjusted life year (QALY) gained will be calculated to assess cost effectiveness.
Difference in HRQOL scores between the treatment groups | 3, 7 weeks post-surgery; 6 months post-surgery; 1, 1.5, 2, 3, 4, 5 years post-surgery
  Difference in HRQOL scores between the treatment groups, as measured by the EQ-5D-5L questionnaire at weeks 3 and 7; months 6, 12, 18, 24; and years 3, 4, and 5, which coincide with the intervals of oncological surveillance.
Difference in 5-year survival rate between the two groups | 5 years post-surgery
  Difference in 5-year survival rate between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Waël C Hanna, MDCM, MBA, FRCSC, Principal Investigator — McMaster University
Locations (1):
- McMaster University / St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grogan EL, Jones DR. VATS lobectomy is better than open thoracotomy: what is the evidence for short-term outcomes? Thorac Surg Clin. 2008 Aug;18(3):249-58. doi: 10.1016/j.thorsurg.2008.04.007. PMID 18831499
- [Background] Onaitis MW, Petersen RP, Balderson SS, et al. Thoracoscopic Lobectomy Is a Safe and Versatile Procedure. Transactions of the Meeting of the American Surgical Association. 2006;124:86-91. doi:10.1097/01.sla.0000234892.79056.63.
- [Background] Veronesi G. Robotic thoracic surgery: technical considerations and learning curve for pulmonary resection. Thorac Surg Clin. 2014 May;24(2):135-41, v. doi: 10.1016/j.thorsurg.2014.02.009. PMID 24780416
- [Background] Nasir BS, Bryant AS, Minnich DJ, Wei B, Cerfolio RJ. Performing robotic lobectomy and segmentectomy: cost, profitability, and outcomes. Ann Thorac Surg. 2014 Jul;98(1):203-8; discussion 208-9. doi: 10.1016/j.athoracsur.2014.02.051. Epub 2014 May 1. PMID 24793685
- [Background] Park BJ, Melfi F, Mussi A, Maisonneuve P, Spaggiari L, Da Silva RK, Veronesi G. Robotic lobectomy for non-small cell lung cancer (NSCLC): long-term oncologic results. J Thorac Cardiovasc Surg. 2012 Feb;143(2):383-9. doi: 10.1016/j.jtcvs.2011.10.055. Epub 2011 Nov 20. PMID 22104677
- [Background] Wei B, D'Amico TA. Thoracoscopic versus robotic approaches: advantages and disadvantages. Thorac Surg Clin. 2014 May;24(2):177-88, vi. doi: 10.1016/j.thorsurg.2014.02.001. PMID 24780422
- [Background] Louie BE, Farivar AS, Aye RW, Vallieres E. Early experience with robotic lung resection results in similar operative outcomes and morbidity when compared with matched video-assisted thoracoscopic surgery cases. Ann Thorac Surg. 2012 May;93(5):1598-604; discussion 1604-5. doi: 10.1016/j.athoracsur.2012.01.067. Epub 2012 Mar 20. PMID 22440364
- [Background] Kent M, Wang T, Whyte R, Curran T, Flores R, Gangadharan S. Open, video-assisted thoracic surgery, and robotic lobectomy: review of a national database. Ann Thorac Surg. 2014 Jan;97(1):236-42; discussion 242-4. doi: 10.1016/j.athoracsur.2013.07.117. Epub 2013 Oct 1. PMID 24090577
- [Background] Paul S, Jalbert J, Isaacs AJ, Altorki NK, Isom OW, Sedrakyan A. Comparative effectiveness of robotic-assisted vs thoracoscopic lobectomy. Chest. 2014 Dec;146(6):1505-1512. doi: 10.1378/chest.13-3032. PMID 24810546
- [Background] Hanna, WC., Fahim, C., Patel, P., Shargall, Y., Waddell TK., Yasufuku, K. (2015). Robotic Pulmonary Resection for Lung Cancer: The First Canadian Series. Abstract Accepted for podium presentation at Canadian Association of Thoracic Surgeons (CATS) 18th Annual Meeting, September 17-20, Quebec, QC.
- [Background] Merritt RE, Hoang CD, Shrager JB. Lymph node evaluation achieved by open lobectomy compared with thoracoscopic lobectomy for N0 lung cancer. Ann Thorac Surg. 2013 Oct;96(4):1171-1177. doi: 10.1016/j.athoracsur.2013.05.044. Epub 2013 Jul 31. PMID 23915591
- [Background] D'Amico TA, Niland J, Mamet R, Zornosa C, Dexter EU, Onaitis MW. Efficacy of mediastinal lymph node dissection during lobectomy for lung cancer by thoracoscopy and thoracotomy. Ann Thorac Surg. 2011 Jul;92(1):226-31; discussion 231-2. doi: 10.1016/j.athoracsur.2011.03.134. PMID 21718849
- [Background] Research Electronic Data Capture (RedCap). http://www.project-redcap.org
- [Background] Cerfolio RJ. Total port approach for robotic lobectomy. Thorac Surg Clin. 2014 May;24(2):151-6, v. doi: 10.1016/j.thorsurg.2014.02.006. PMID 24780418
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Cerfolio RJ, Bryant AS. How to teach robotic pulmonary resection. Semin Thorac Cardiovasc Surg. 2013 Spring;25(1):76-82. doi: 10.1053/j.semtcvs.2013.01.004. No abstract available. PMID 23800532
- [Background] Pickard AS, Neary MP, Cella D. Estimation of minimally important differences in EQ-5D utility and VAS scores in cancer. Health Qual Life Outcomes. 2007 Dec 21;5:70. doi: 10.1186/1477-7525-5-70. PMID 18154669
- [Background] Little, R.J.A. and Rubin, D.B. (1987) Statistical Analysis with Missing Data. J. Wiley & Sons, New York.
- [Background] SAS Institute Inc., SAS 9.4 Help and Documentation, Cary, NC: SAS Institute Inc., 2000-2012.
- [Derived] Patel YS, Hanna WC, Fahim C, Shargall Y, Waddell TK, Yasufuku K, Machuca TN, Pipkin M, Baste JM, Xie F, Shiwcharan A, Foster G, Thabane L. RAVAL trial: Protocol of an international, multi-centered, blinded, randomized controlled trial comparing robotic-assisted versus video-assisted lobectomy for early-stage lung cancer. PLoS One. 2022 Feb 2;17(2):e0261767. doi: 10.1371/journal.pone.0261767. eCollection 2022. PMID 35108265
- [Derived] Ujiie H, Gregor A, Yasufuku K. Minimally invasive surgical approaches for lung cancer. Expert Rev Respir Med. 2019 Jun;13(6):571-578. doi: 10.1080/17476348.2019.1610399. Epub 2019 May 6. PMID 31055977